CLINICAL TRIAL: NCT04455477
Title: Hemodynamic Effects of Nesiritide on Congestive Heart Failure Patients Receiving Mechanical Ventilation: A Prospective Observational Study
Brief Title: Nesiritide for Ventilated Congestive Heart Failure
Acronym: HENCHF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2020-056R
Record Dates: First submitted 2020-05-16; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Congestive Heart Failure; Mechanical Ventilation; Using Nesiritide; Venous Return; Cardiac Function
Keywords: Congestive Heart Failure; Nesiritide
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Nesiritide — The attending physicans decide whether to use Nesiritide for congestive heart failure patients. Only patients who will use Nesiritide are enrolled.

SUMMARY:
The congestive heart failure is a common disease among patients who receive cardiac surgery and may lead to prolonged ventilation support. Nesiritide was a potential therapy for congestive heart failure. This study aimed to compare the Nesiritide induced hemodynamical status changes among congestive heart failure patients with invasive ventilation support.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years；
* Congestive Heart Failure;
* With mechanical ventilation；
* With hemodynamic monitoring devices;
* The physicians made the decision of using Nesiritide.

Exclusion Criteria:

* Unstable hemodynamic status；
* Severe renal dysfunction.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Congestive heart failure patients relying on mechanical ventilation and therefore decide to try the Nesiritide.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of cardiac output | Before and 30-min after using a standard dose of Nesiritide
  Changes of cardiac output measured by hemodynamical monitoring tools
Changes of systemic filling pressure | Before and 30-min after using a standard dose of Nesiritide
  Changes of the intercept of regression line of paired VR-RAP points at different PEEP levels.

SECONDARY OUTCOMES:
Changes of cardiac function curve | Before and 30-min after using a standard dose of Nesiritide
  Using body position changes (±15°) to simulate the change of preload, and therefore depicte the Starling curve
Changes of venous return curve | Before and 30-min after using a standard dose of Nesiritide
  Changes of venous return curve depicted by different PEEP setting

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Xuhui, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Our institution did not approve this.